CLINICAL TRIAL: NCT02476708
Title: A Pilot Trial of Curcumin Effects on Cognition in Schizophrenia
Acronym: CRC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was not achieved as expected
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Cenk Tek, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1412015121
Record Dates: First submitted 2015-05-05; First posted 2015-06-19 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; cognition; curcumin
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curcumin 1800mg (Experimental): curcumin capsule 600mg taken 3 times per day for 8 weeks
  Interventions: Dietary Supplement: curcumin 1800mg
- Placebo (Placebo Comparator): placebo capsule taken 3 times per day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: curcumin 1800mg — Curcumin, derived from turmeric root, is an over-the-counter supplement which is tolerated well.
  Other Names: theracurmin
  Arms: Curcumin 1800mg
Dietary Supplement: Placebo — oral placebo capsule
  Arms: Placebo

SUMMARY:
This is an 8-week randomized, double-blind, placebo-controlled, parallel, fixed-dose pilot clinical trial of curcumin for the treatment of cognitive impairment in schizophrenia.The primary aim of this pilot trial is to provide an effect size estimate for the efficacy of curcumin in improving cognitive functioning in schizophrenia. Secondary goals are to determine the effect of curcumin over time on negative and positive symptoms, in association with inflammatory markers.

DETAILED DESCRIPTION:
This is an 8-week randomized, double-blind, placebo-controlled, parallel, fixed-dose pilot clinical trial of curcumin for the treatment of cognitive impairment in schizophrenia. Cognitive impairment and persistent negative symptoms are the core dimensions of schizophrenia; however current antipsychotic treatment fails to address this issue. Evidence suggests cognitive impairment is not only limited to patients with late-stage schizophrenia. High rates of cognitive impairment in patients with first episode psychosis indicate that cognitive impairment is not solely a consequence of long-term antipsychotic treatment, but rather is an enduring problem over the course of schizophrenia. Likewise, negative symptoms persist throughout its entire course, and are associated with poor overall functioning. Currently, there are no pharmacological agents that specifically aim to treat cognitive functioning and persistent negative symptoms; therefore, there is growing interest in the development of effective treatments for this unmet need.

The primary aim of this pilot trial is to provide an effect size estimate for the efficacy of curcumin in improving cognitive functioning in schizophrenia. Secondary goals are to determine the effect of curcumin over time on negative and positive symptoms, in association with inflammatory markers. Eligible participants will be randomized to curcumin (n=20) or placebo (n=20) in a 1:1 ratio. A commercially available surface-controlled water soluble form of 600mg curcumin (10% formulation) or matching placebo capsules will be administered three times a day for a total of 8 weeks.

ELIGIBILITY:
Inclusion criteria:

1. 18 - 65 years of age
2. English speaking
3. Diagnostic and Statistical Manual- IV diagnosis of schizophrenia or schizoaffective disorder based on Structured Clinical Interview for Diagnostic and Statistical Manual-IV (SCID)
4. Symptomatic stability confirmed by clinical staff in the 8 weeks prior to the study
5. No changes in antipsychotic medication within the last 8 weeks
6. No change in antipsychotic dose in in last 4 weeks.

Exclusion criteria are:

1. Unable to provide informed consent
2. Diagnostic and Statistical Manual-IV (DSM-IV) diagnosis of alcohol/substance dependence
3. Recent history of gastrointestinal bleeding or ulceration
4. Recent history of gallstones and/or bile duct obstruction
5. Significant uncontrolled systemic illness (e.g. chronic renal failure, chronic liver disease, poorly controlled diabetes, poorly controlled congestive heart failure, chronic infectious disease, chronic autoimmune disease)
6. Known intolerance to turmeric, curcumin, or curry
7. Pregnancy or breast-feeding
8. Current use of anti-platelet, anti-coagulant, glucocorticoid, immunosuppressants
9. Daily use of non-steroidal anti-inflammatory use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Efficacy of curcumin (MATRICS - Composite Score t score) | 8 weeks
  The primary outcome will estimate the efficacy of curcumin in improving cognitive functioning in schizophrenia. This would be measured by comparing change in cognition scores (MATRICS Consensus Cognitive Battery Composite Score) between baseline and endpoint based on medication assignment.

SECONDARY OUTCOMES:
Effect on psychiatric symptoms (PANSS - Positive Score) | 8 weeks
  Secondary outcome will be the effect of curcumin over time on negative and positive symptoms. This will be measured by comparing change in scores on PANSS (Positive and Negative Symptom Scale - Positive Symptom Score 7 min, 49 max) between baseline and endpoint based on medication assignment.
Effect on psychiatric symptoms (PANSS- Negative Score) | 8 weeks
  Secondary aim is to determine the effect of curcumin over time on negative and positive symptoms. This will be measured by comparing change in scores on PANSS (Positive and Negative Symptom Scale - Negative Symptom Score - 7 min, 49 max) between baseline and endpoint based on medication assignment.
Effect on psychiatric symptoms (PANSS- Total Score) | 8 weeks
  Secondary aim is to determine the effect of curcumin over time on negative and positive symptoms. This will be measured by comparing change in scores on PANSS (Positive and Negative Symptom Scale - Total score 14 min, 112 max) between baseline and endpoint based on medication assignment.
Efficacy of curcumin (MATRICS - Speed of Processing - t score) | 8 weeks
  This outcome will estimate the efficacy of curcumin in improving cognitive functioning in schizophrenia. This would be measured by comparing change in cognition scores. MATRICS Consensus Cognitive Battery Speed of Processing is calculated from the composite of t-scores for trail making task (time in seconds - max 300), Brief Assessment of Cognition in Schizophrenia (number of correct responses, max 110), and fluency/animal naming (number of animals named in 60 seconds) between baseline and endpoint based on medication assignment.
Efficacy of curcumin (MATRICS - Attention/Vigilance t-score) | 8 weeks
  This outcome will estimate the efficacy of curcumin in improving cognitive functioning in schizophrenia. This would be measured by comparing change in cognition scores. MATRICS Consensus Cognitive Battery Attention/Vigilance is calculated as the computer-generated score from the Continuous Performance Test - Identical Pairs (CPT-IP) program between baseline and endpoint based on medication assignment.
Efficacy of curcumin (MATRICS - Working Memory t-score) | 8 weeks
  This outcome will estimate the efficacy of curcumin in improving cognitive functioning in schizophrenia. This would be measured by comparing change in cognition scores. MATRICS Consensus Cognitive Battery Working Memory is calculated from the composite of t-scores for the Wechsler Memory Scale-III: Spacial Span (Sum of forward and backward total scores, range 0-32) between baseline and endpoint based on medication assignment.
Efficacy of curcumin (MATRICS - Verbal Learning t-score) | 8 weeks
  This outcome will estimate the efficacy of curcumin in improving cognitive functioning in schizophrenia. This would be measured by comparing change in cognition scores. MATRICS Consensus Cognitive Battery Verbal Learning is calculated as the total number of words recalled from the Hopkins-Verbal Learning Test-revised (range 0-36) between baseline and endpoint based on medication assignment.
Efficacy of curcumin (MATRICS - Visual Learning t-score) | 8 weeks
  This outcome will estimate the efficacy of curcumin in improving cognitive functioning in schizophrenia. This would be measured by comparing change in cognition scores. MATRICS Consensus Cognitive Battery Visual Learning is calculated as the total score from the Brief Visuospacial Memory Test - revised (range 0-36) between baseline and endpoint based on medication assignment.
Efficacy of curcumin (MATRICS - Reasoning and Problem Solving t-score) | 8 weeks
  This outcome will estimate the efficacy of curcumin in improving cognitive functioning in schizophrenia. This would be measured by comparing change in cognition scores. MATRICS Consensus Cognitive Battery Reasoning and Problem Solving is calculated as the total score for the 7 mazes as part of the Neuropsychological Assessment Battery (NAB) mazes (range 0-26) between baseline and endpoint based on medication assignment.
Efficacy of curcumin (MATRICS - Social Cognition t-score) | 8 weeks
  This outcome will estimate the efficacy of curcumin in improving cognitive functioning in schizophrenia. This would be measured by comparing change in cognition scores. MATRICS Consensus Cognitive Battery Social Cognition is a computer generated branch score calculated from performance on the Mayer-Salovey-Caruso Emotional Intellegence Test (MSCEIT): Managing Emotions between baseline and endpoint based on medication assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Tek, MD, Principal Investigator — Yale Unversity School of Medicine
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data resulting from this award involving human subjects will be submitted to the NIMH Data Archive (NDA) - National Database for Clinical Trials Related to Mental Illness (NDCT) The Principal Investigator will work with NDA support staff to plan an appropriate data submission schedule and provide information on the steps for submission and sharing of data. Communication of this data sharing plan to appropriate research staff to ensure the timely submission of data. All human subject data provided will include an NDA Global Unique Identifier (GUID) and will not include personally identifiable information (PII). Analyzed data will be submitted no later than the time of publication. Even if a publication focuses on only part of an analyzed dataset, the entire analyzed dataset will be submitted when the first paper is published. All data made available for public use via NDA will be de-identified data.